CLINICAL TRIAL: NCT03411863
Title: Noninvasive Cervical Electrical Stimulation for ALS: Mechanistic and Safety Study
Brief Title: Cervical Electrical Stimulation for ALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: B2527-P
Record Dates: First submitted 2018-01-05; First posted 2018-01-26 (Actual); Results first posted 2022-10-25 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-09

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Transcutaneous Electric Nerve Stimulation; transcranial magnetic stimulation
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Participants without neurological disease (Active Comparator): Participants without neurological disease. All subjects undergo the same full protocol.
  Interventions: Device: CES at rest; Device: CES plus active hand or wrist movements
- Participants with ALS (Experimental): Participants with ALS. All subjects undergo the same full protocol.
  Interventions: Device: CES at rest; Device: CES plus active hand or wrist movements

INTERVENTIONS:
Device: CES at rest — CES will be delivered at rest at various intensities, in combination with either electrical stimulation over peripheral nerves or magnetic stimulation over the motor cortex.
  This is an experiment designed to measure CES interactions with other central and peripheral nerve circuits.
Device: CES plus active hand or wrist movements — CES will be delivered while the participant performs specific finger or wrist tasks at different degrees of effort.
  This is an experiment designed to detect momentary changes in muscle function.

SUMMARY:
Veterans are at higher risk than non-Veterans of falling ill with amyotrophic lateral sclerosis (ALS). ALS causes degeneration of motor neurons in both the brain and the spinal cord. Evidence from studies in people with spinal cord injury suggests that activating spared nerve circuits with electromagnetic stimulation improves nerve transmission.

With this goal, the investigators have developed a novel method of noninvasive cervical (neck) electrical stimulation (CES). In this study, the investigators will investigate CES for its potential to strengthen nerve circuits to the hands in ALS.

To the investigators' knowledge, electrical spinal stimulation for ALS has never been tested previously. This study will be performed in two stages: First, basic experiments will be performed to better understand how CES interacts with other types of electrical and magnetic stimulations over the brain and peripheral nerves. Second, experiments will be performed to determine the types of CES that can facilitate active arm and hand movements.

These experiments will improve understanding of electrical stimulation in ALS, and may set the table for future treatments.

Both United States Veterans and non-Veterans are eligible to participate in this study.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) reduces connections between the cortical motor neurons that initiate movement and the spinal motor neurons that direct muscles to execute movement. This situation shares many key features with incomplete spinal cord injury (SCI). Accumulating evidence in SCI suggests that externally activating spared nerve circuits with electromagnetic stimulation augments neural transmission.

With this goal, the investigators developed a novel method of noninvasive cervical electrical stimulation (CES). CES activates multiple muscles on both upper limbs by triggering afferent sensory or efferent motor nerve roots depending on stimulus intensity. This study will investigate CES for its potential to strengthen residual circuits to the hands in ALS.

To the investigators' knowledge, electrical spinal stimulation for ALS has never been tested or applied previously. Therefore, a pilot study is essential. This study will be performed in two stages:

1. Map CES circuit and synaptic targets: The experiments share a common structure comprising conditioning and test stimuli delivered at a range of intensities, sites, and interstimulus intervals.
2. Determine parameters for combining CES with volitional movement: volitional limb movements depend on the same corticospinal and motor neuron circuits as those activated by TMS and F-waves. Since preliminary data shows that subthreshold CES facilitates transcranial magnetic stimulation (TMS) responses, CES may also be able to facilitate volitional limb movements.

Successful completion of these experiments will: mechanistically elucidate CES circuit interactions; investigate the potential for CES to enhance concurrent volitional muscle activation; and establish CES as safe and feasible in the ALS population. Given the limited treatment options for ALS, any amount of progress would represent a meaningful step forward. Moreover, results of this pilot study could lead to direct translation for lasting clinical benefit by combining repetitive subthreshold CES with repetitive task-oriented physical exercise training in subsequent studies. CES would be compatible with other interventions, including medications and cell-based treatments.

ELIGIBILITY:
Inclusion Criteria (ALS):

* Age between 21 and 75 years
* Diagnosis of probable or definite ALS (or non-disabled volunteer)
* Incomplete weakness of left or right wrist or hand muscles:

  * score of 2, 3, or 4 (out of 5) on manual muscle testing of:
  * wrist flexion
  * finger extension
  * finger flexion
  * or finger abduction
* Detectable F-wave responses of the left or right abductor pollicis brevis (APB) to median nerve stimulation and/or adductor digiti minimi (ADM) to ulnar nerve stimulation
* US Veteran or non-Veteran

Inclusion Criteria (Participants without neurological disease):

* Age between 21 and 75 years
* No history of significant neurological disease
* Detectable F-wave responses of the left or right APB to median nerve stimulation and/or ADM to ulnar nerve stimulation
* US Veteran or non-Veteran

Exclusion Criteria (ALS):

* History of other serious injury or disease of central or peripheral nervous system
* History of seizures
* Ventilator dependence or patent tracheostomy site
* Use of medications that significantly lower seizure threshold
* History of head trauma with evidence of brain contusion or hemorrhage or depressed skull fracture on prior imaging
* History of implanted:

  * brain/spine/nerve stimulators
  * aneurysm clips
  * ferromagnetic metallic implants
  * or cardiac pacemaker/defibrillator
* Significant coronary artery or cardiac conduction disease
* History of bipolar disorder or suicide attempt or active psychosis
* Heavy alcohol consumption (> equivalent of 5 oz of liquor) within previous 48 hours
* Open skin lesions over the face, neck, shoulders, or arms
* Pregnancy
* Unsuitable for study participation as determined by study physician

Exclusion Criteria: (Participants without neurological disease)

* History of other serious injury or disease of central or peripheral nervous system
* History of seizures
* Ventilator dependence or patent tracheostomy site
* Use of medications that significantly lower seizure threshold
* History of head trauma with evidence of brain contusion or hemorrhage or depressed skull fracture on prior imaging
* History of implanted:

  * brain/spine/nerve stimulators
  * aneurysm clips
  * ferromagnetic metallic implants
  * or cardiac pacemaker/defibrillator
* Significant coronary artery or cardiac conduction disease
* History of bipolar disorder or suicide attempt or active psychosis
* Heavy alcohol consumption (> equivalent of 5 oz of liquor) within previous 48 hours
* Open skin lesions over the face, neck, shoulders, or arms
* Pregnancy
* Unsuitable for study participation as determined by study physician

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noam Y. Harel, MD PhD, Principal Investigator — James J. Peters Veterans Affairs Medical Center
Locations (1):
- James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
A Limited Dataset (LDS), with individual electrophysiological and physiological outcome measures, will be shared in electronic format pursuant to a VA-approved Data Use Agreement. Individually Identifiable Data will be shared pursuant to valid HIPAA Authorization, Informed Consent, and an appropriate written agreement limiting use of the data to the conditions as described in the authorization and consent, and a written assurance from the recipient that the information will be maintained in accordance with the security requirements of 38 Code of Federal Regulations (CFR) Part 1.466.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At time of publication.
Access Criteria: A Limited Dataset (LDS) will be shared in electronic format pursuant to a VA-approved Data Use Agreement. Individually Identifiable Data will be shared pursuant to valid HIPAA Authorization, Informed Consent, and an appropriate written agreement limiting use of the data to the conditions as described in the authorization and consent, and a written assurance from the recipient that the information will be maintained in accordance with the security requirements of 38 CFR Part 1.466.

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants Without Neurological Disease; Participants With Amyotrophic Lateral Sclerosis (ALS): All subjects undergo same full protocol.
  CES at rest: CES will be delivered at rest at various intensities, in combination with either electrical stimulation over peripheral nerves or magnetic stimulation over the motor cortex.
  This is an experiment designed to measure CES interactions with other central and peripheral nerve circuits.
  CES plus active hand or wrist movements: CES will be delivered while the participant performs specific finger or wrist tasks at different degrees of effort.
  This is an experiment designed to detect momentary changes in muscle function.
Period: Overall Study
Arm/Group | Participants Without Neurological Disease | Participants With Amyotrophic Lateral Sclerosis (ALS)
Started | 8 | 11
Completed | 5 | 9
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Participants With ALS: All subjects undergo same full protocol.
  CES at rest: CES will be delivered at rest at various intensities, in combination with either electrical stimulation over peripheral nerves or magnetic stimulation over the motor cortex.
  This is an experiment designed to measure CES interactions with other central and peripheral nerve circuits.
  CES plus active hand or wrist movements: CES will be delivered while the participant performs specific finger or wrist tasks at different degrees of effort.
  This is an experiment designed to detect momentary changes in muscle function.
- Total: Total of all reporting groups
Arm/Group | Participants Without Neurological Disease | Participants With ALS | Total
Number analyzed (Participants) | 8 | 11 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 10 | 17
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 5 | 6 | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 11 | 19

OUTCOME MEASURES:

1. Primary Outcome: Electromyographic (EMG) Responses (Rest)
Description: These results are derived from peak-to-peak EMG amplitude in the abductor pollicis brevis (APB) muscle in response to transcranial magnetic stimulation (TMS). Values represent the ratio of peak-to-peak APB amplitude when TMS is paired with cervical electrical stimulation (CES) at the indicated timing (in milliseconds) normalized to the response to TMS alone (control).
Time Frame: up to 1 day
Population: Participants who completed at least one session of resting conditioned/non-conditioned stimuli were analyzed.
Measure: Mean (Standard Deviation); unit: % change compared to TMS alone
Groups:
- Participants Without Neurological Disease: Participants without neurological disease.
- Participants With Amyotrophic Lateral Sclerosis (ALS): Participants with ALS.
Arm/Group | Participants Without Neurological Disease | Participants With Amyotrophic Lateral Sclerosis (ALS)
Number analyzed (Participants) | 6 | 7
% change compared to TMS alone
  TMS+CES -25 ms | 6.8 (29.0) | 21.6 (44.7)
  TMS+CES -10 ms | 8.4 (25.5) | -6.1 (17.9)
  TMS+CES -2 ms | 8.0 (24.9) | 3.4 (42.0)
  TMS+CES 0 ms | 2.7 (53.2) | 38.5 (38.6)
  TMS+CES +2 ms | -5.9 (23.6) | 48.3 (67.2)
  TMS+CES +5 ms | 14.1 (38.7) | 11.2 (39.0)
  TMS+CES +10 ms | 14.0 (30.4) | 45.8 (77.0)

2. Primary Outcome: Electromyographic Responses (Active)
Description: Effect of CES on concurrent finger or wrist active movements will be measured via root-mean-square of ongoing muscle activity in various hand and forearm muscles.
Time Frame: up to 1 day
Population: Unfortunately, this data is uninterpretable due to technically mis-timed synchronization between muscle action and spinal stimulation.
Groups:
- Participants With ALS: Participants with ALS.
Arm/Group | Participants Without Neurological Disease | Participants With ALS
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 hours
Groups:
- Participants Without Neurological Injury; Participants With ALS: All subjects undergo same full protocol.
  CES at rest: CES will be delivered at rest at various intensities, in combination with either electrical stimulation over peripheral nerves or magnetic stimulation over the motor cortex.
  This is an experiment designed to measure CES interactions with other central and peripheral nerve circuits.
  CES plus active hand or wrist movements: CES will be delivered while the participant performs specific finger or wrist tasks at different degrees of effort.
  This is an experiment designed to detect momentary changes in muscle function.
Arm/Group | Participants Without Neurological Injury | Participants With ALS
All-Cause Mortality (participants affected / at risk) | 0/8 | 5/11
Serious Adverse Events (participants affected / at risk) | 0/8 | 1/11
Other Adverse Events (participants affected / at risk) | 2/8 | 5/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Without Neurological Injury (N=8) | Participants With ALS (N=11)
Unrelated hand laceration (Injury, poisoning and procedural complications) | 0 | 1 (1) — Participant suffered hand laceration requiring emergency department visit and sutures while working in his home workshop. Unrelated to study procedures.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Without Neurological Injury (N=8) | Participants With ALS (N=11)
Headache (Nervous system disorders) | 1 (1) | 4 (4)
Flushing (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (5)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Sore throat (Gastrointestinal disorders) | 0 (0) | 1 (2)
Blurry vision (Eye disorders) | 0 (0) | 1 (1) — less than 1 second
Light-headed (Nervous system disorders) | 1 (1) | 0 (0)
Metallic taste (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-05): https://cdn.clinicaltrials.gov/large-docs/63/NCT03411863/Prot_SAP_000.pdf